CLINICAL TRIAL: NCT04789694
Title: Prehabilitation in Patients With Gynaecological Cancer Planned for Postponed Surgical Management: A Prospective Randomised Trial.
Brief Title: Prehabilitation in Gynaecological Cancer Patients
Acronym: PHOCUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University Hospital Ostrava (Other); University Hospital Olomouc (Other); University Hospital Pilsen (Other); The Faculty Hospital Na Bulovce (Other)
Responsible Party: Principal Investigator, David Cibula, professor, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHOCUS_38/20
Record Dates: First submitted 2021-02-01; First posted 2021-03-09 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer; Ovarian Cancer Stage III; Ovarian Cancer Stage IV; Endometrial Cancer; Frailty
Keywords: Prehabilitation; Epitelial ovarian cancer; Functional capacity; Quality of life; Multimodal prehabilitation; Frailty; Endometrial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Frailty | interventions — Psychosocial Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (No Intervention): Patients will be provided with a basic information and standard of care support.
- B (Experimental): Active prehabilitation will be provided, composed of i) three physical activity-related interventions provided by a physical and rehabilitation medicine (PRM) specialist; iii) three 30 min consultations regarding nutritional status with physician or nutrition specialist; ii) three sessions with psychologist.
  Interventions: Other: Physiological intervention; Behavioral: Psychological intervention; Dietary Supplement: Nutritional intervention

INTERVENTIONS:
Other: Physiological intervention — * Rehabilitation specialist consultation (3x)
  * Individualized home-based exercise plan
  * Functional capacity measuring
  Arms: B
Behavioral: Psychological intervention — * Clinical psychologist consultation (3x)
  * Anxiety and depression scoring
  * Psychological support
  Arms: B
Dietary Supplement: Nutritional intervention — * Nutritional specialist consultation (3x)
  * Malnutrition scoring
  * Dietary supplementation
  Arms: B

SUMMARY:
Prehabilitation refers to interventions aiming to improve patients' resilience and functional capacity before a known stressful event, e.g., scheduled surgery. These interventions usually consist of physical activity and psychological and nutritional support. There is substantial evidence of the positive effect of multimodal prehabilitation among patients treated surgically for non-gynaecological cancers; however, no prospective data are available in gynaecological cancer patients.

PHOCUS trial is a prospective randomised trial aiming to evaluate the role of multimodal prehabilitation in patients with gynaecological cancer. Sixty-four patients will be randomised in single institution within 36 months with a 1:1 ratio into ARM A: control arm which will be provided with a basic information and standard of care support; ARM B: active arm undergoing multimodal prehabilitation composed of physical activity and psychological and nutritional support. All patients will be assessed at standard intervals (three times during the trial) by a spectrum of non-invasive tests, evaluating physical functional capacity, postoperative morbidity, nutritional status, level of stress and anxiety, and quality of life.

DETAILED DESCRIPTION:
The objective of the trial is to evaluate the impact of intensive multimodal prehabilitation protocol on pre-operative functional capacity, postoperative morbidity, and quality of life in patients undergoing surgical treatment for gynaecological cancer.

Two groups of patients scheduled for postponed surgical treatment will be eligible for the trial: i) advanced ovarian cancer patients referred for neoadjuvant chemotherapy and interval debulking surgery; ii) stage I-II endometrial cancer patients classifying as frail (according to the validated modified Frailty Index), who will be treated by hormonal therapy for three months, followed by surgical treatment.

ELIGIBILITY:
Inclusion criteria

Two groups of patients will be eligible for the trial:

i) Epithelial ovarian cancer patients referred for NACT: a) FIGO stage III or IV disease; b) Patient is not a candidate for primary debulking surgery; c) Patient is a suitable candidate for standard of care combined chemotherapy; d) Patient is a candidate for interval.debulking surgery

ii) Stage I or II endometrial cancer patients classifying as frail according to the validated modified Frailty Index: a) FIGO stage I or II; b) Patient is classified as frail; c) Patient is suitable candidate for hormonal therapy.

Exclusion criteria

1. Second malignant tumour (under the treatment)
2. Patient is not suitable for any surgery delay
3. Patient is not physically able to meet the prehabilitation intervention plan or is unable to walk

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Functional capacity changes | 9-12weeks
  Six-minute walking test (6MWT)

SECONDARY OUTCOMES:
Postoperative morbidity | 9-12weeks
  Intraoperative and early postoperative complications until the 30th postoperative day will be classified according to the Clavien-Dindo and the Comprehensive Complication Index. Adverse events occurring after 30th postoperative day will be assessed according to NCI Common Terminology Criteria for Adverse Events Version 5.0
Length of postoperative hospital stay (days) | 9-12weeks
Adherence to training program | 9-12weeks
  Daily step count and number of resistance exercises per week.
Effects of nutritional support program on body composition (weight of fat and lean body mass in kg) | 9-12weeks
Effects of nutritional support program on resting energy expenditure (measured in kcal/kg). | 9-12weeks
Effects of nutritional support program on Fatty acids composition of plasmatic and erythrocytes phospholipids (measured in mol%). | 9-12weeks
Health-related quality of life | 9-12weeks
  The analysis of the QoL of both study ARMs will be made based on EORTC validated questionnaires: QLQ-C30 and OV28 (for ovarian cancer patients)/ EN24 (for endometrial cancer patients.
  QLQ-C30 was developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials. The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  The EORTC QLQ-OV28/ EN24 is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 25 items specifically related to ovarian/ endometrial cancer.
Psychological health: DEPRESSION | 9-12weeks
  The Beck Depression Inventory: a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.
Psychological health: ANXIETY | 9-12weeks
  The State-Trait Anxiety Inventory: a psychological inventory consisting of 40 self-report items on a 4-point Likert scale. The STAI measures two types of anxiety - state anxiety and trait anxiety.
Psychological health: NONSPECIFIC PERCEIVED STRESS | 9-12weeks
  Perceived stress scale: psychological instrument for measuring nonspecific perceived stress (stressfulness of situations, the effectiveness of stress-reducing interventions, and the extent to which there are associations between psychological stress and psychiatric and physical disorders).
Psychological health: SPECIFIC PERCEIVED STRESS | 9-12weeks
  Stress profile: questionnaire assessing the severity of stress in nine areas of life: social habits, social relationships, life events, sexual problems, sleep, psychiatric symptoms, old age, menstrual stresses, and 'stress and the heart'.

CONTACTS AND LOCATIONS:
Overall Officials: David Cibula, prof., Principal Investigator — Charles University, Czech Republic
Locations (1):
- Gynecologic Oncology Center in Prague, Prague, Czechia

REFERENCES:
- [Background] Cook PC, Leit ME. Issues in the pediatric athlete. Orthop Clin North Am. 1995 Jul;26(3):453-64. PMID 7609960
- [Background] Althoff FC, Neb H, Herrmann E, Trentino KM, Vernich L, Fullenbach C, Freedman J, Waters JH, Farmer S, Leahy MF, Zacharowski K, Meybohm P, Choorapoikayil S. Multimodal Patient Blood Management Program Based on a Three-pillar Strategy: A Systematic Review and Meta-analysis. Ann Surg. 2019 May;269(5):794-804. doi: 10.1097/SLA.0000000000003095. PMID 30418206
- [Background] Peteroy ET, Pirrello PE, Adams N. The relationship between two Wiggins Content Scales and length of hospitalization. J Clin Psychol. 1982 Apr;38(2):344-6. doi: 10.1002/1097-4679(198204)38:23.0.co;2-z. PMID 7068871
- [Background] Barberan-Garcia A, Ubre M, Roca J, Lacy AM, Burgos F, Risco R, Momblan D, Balust J, Blanco I, Martinez-Palli G. Personalised Prehabilitation in High-risk Patients Undergoing Elective Major Abdominal Surgery: A Randomized Blinded Controlled Trial. Ann Surg. 2018 Jan;267(1):50-56. doi: 10.1097/SLA.0000000000002293. PMID 28489682
- [Background] Beck A, Vind Thaysen H, Hasselholt Soegaard C, Blaakaer J, Seibaek L. Prehabilitation in cancer care: patients' ability to prepare for major abdominal surgery. Scand J Caring Sci. 2021 Mar;35(1):143-155. doi: 10.1111/scs.12828. Epub 2020 Feb 11. PMID 32043644
- [Background] Benzo R, Wigle D, Novotny P, Wetzstein M, Nichols F, Shen RK, Cassivi S, Deschamps C. Preoperative pulmonary rehabilitation before lung cancer resection: results from two randomized studies. Lung Cancer. 2011 Dec;74(3):441-5. doi: 10.1016/j.lungcan.2011.05.011. Epub 2011 Jun 12. PMID 21663994
- [Background] Biglia N, Zanfagnin V, Daniele A, Robba E, Bounous VE. Lower Body Lymphedema in Patients with Gynecologic Cancer. Anticancer Res. 2017 Aug;37(8):4005-4015. doi: 10.21873/anticanres.11785. PMID 28739682
- [Background] Blackwell JEM, Doleman B, Boereboom CL, Morton A, Williams S, Atherton P, Smith K, Williams JP, Phillips BE, Lund JN. High-intensity interval training produces a significant improvement in fitness in less than 31 days before surgery for urological cancer: a randomised control trial. Prostate Cancer Prostatic Dis. 2020 Dec;23(4):696-704. doi: 10.1038/s41391-020-0219-1. Epub 2020 Mar 10. PMID 32157250
- [Background] Burden S, Todd C, Hill J, Lal S. Pre-operative nutrition support in patients undergoing gastrointestinal surgery. Cochrane Database Syst Rev. 2012 Nov 14;11:CD008879. doi: 10.1002/14651858.CD008879.pub2. PMID 23152265
- [Background] Burke SM, Brunet J, Sabiston CM, Jack S, Grocott MP, West MA. Patients' perceptions of quality of life during active treatment for locally advanced rectal cancer: the importance of preoperative exercise. Support Care Cancer. 2013 Dec;21(12):3345-53. doi: 10.1007/s00520-013-1908-2. Epub 2013 Aug 3. PMID 23912669
- [Background] Carli F, Brown R, Kennepohl S. Prehabilitation to enhance postoperative recovery for an octogenarian following robotic-assisted hysterectomy with endometrial cancer. Can J Anaesth. 2012 Aug;59(8):779-84. doi: 10.1007/s12630-012-9734-4. Epub 2012 May 26. PMID 22638674
- [Background] Cianci S, Tarascio M, Rosati A, Caruso S, Uccella S, Cosentino F, Scaletta G, Gueli Alletti S, Scambia G. Sexual function and quality of life of patients affected by ovarian cancer. Minerva Med. 2019 Aug;110(4):320-329. doi: 10.23736/S0026-4806.19.06080-4. Epub 2019 May 6. PMID 31081305
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Cortes-Guiral D, Mohamed F, Glehen O, Passot G. Prehabilitation of patients undergoing cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) for peritoneal malignancy. Eur J Surg Oncol. 2021 Jan;47(1):60-64. doi: 10.1016/j.ejso.2020.01.032. Epub 2020 Jan 30. PMID 32063398
- [Background] Daroszewski C, Stasiewicz M, Jazwinska-Tarnawska E, Rachwalik A, Mura E, Luboch-Kowal J, Drys A, Bogucki ZA, Brzecka A. Quality of Life in Patients with Advanced Non-Small-Cell Lung Cancer Receiving Palliative Chemotherapy. Adv Exp Med Biol. 2019;1160:11-18. doi: 10.1007/5584_2019_346. PMID 30825114
- [Background] Driver JA, Viswanathan AN. Frailty measure is more predictive of outcomes after curative therapy for endometrial cancer than traditional risk factors in women 60 and older. Gynecol Oncol. 2017 Jun;145(3):526-530. doi: 10.1016/j.ygyno.2017.03.010. Epub 2017 Mar 28. PMID 28359689
- [Background] Ekici U, Ferhatoglu MF. Perioperative and Postoperative Effects of Preoperative Low-Calorie Restrictive Diets on Patients Undergoing Laparoscopic Sleeve Gastrectomy. J Gastrointest Surg. 2020 Feb;24(2):313-319. doi: 10.1007/s11605-019-04157-5. Epub 2019 Feb 20. PMID 30788716
- [Background] Gillis C, Buhler K, Bresee L, Carli F, Gramlich L, Culos-Reed N, Sajobi TT, Fenton TR. Effects of Nutritional Prehabilitation, With and Without Exercise, on Outcomes of Patients Who Undergo Colorectal Surgery: A Systematic Review and Meta-analysis. Gastroenterology. 2018 Aug;155(2):391-410.e4. doi: 10.1053/j.gastro.2018.05.012. Epub 2018 May 8. PMID 29750973
- [Background] Gillis C, Li C, Lee L, Awasthi R, Augustin B, Gamsa A, Liberman AS, Stein B, Charlebois P, Feldman LS, Carli F. Prehabilitation versus rehabilitation: a randomized control trial in patients undergoing colorectal resection for cancer. Anesthesiology. 2014 Nov;121(5):937-47. doi: 10.1097/ALN.0000000000000393. PMID 25076007
- [Background] Goode PS. Efficacy of an assisted low-intensity programme of perioperative pelvic floor muscle training in improving the recovery of continence after radical prostatectomy: a randomized controlled trial. BJU Int. 2012 Oct;110(7):1010-1. doi: 10.1111/j.1464-410X.2012.11451.x. Epub 2012 Aug 22. No abstract available. PMID 22909353
- [Background] Gunderson CC, Fader AN, Carson KA, Bristow RE. Oncologic and reproductive outcomes with progestin therapy in women with endometrial hyperplasia and grade 1 adenocarcinoma: a systematic review. Gynecol Oncol. 2012 May;125(2):477-82. doi: 10.1016/j.ygyno.2012.01.003. Epub 2012 Jan 11. PMID 22245711
- [Background] Handforth C, Clegg A, Young C, Simpkins S, Seymour MT, Selby PJ, Young J. The prevalence and outcomes of frailty in older cancer patients: a systematic review. Ann Oncol. 2015 Jun;26(6):1091-1101. doi: 10.1093/annonc/mdu540. Epub 2014 Nov 17. PMID 25403592
- [Background] Cho BC, Serini J, Zorrilla-Vaca A, Scott MJ, Gehrie EA, Frank SM, Grant MC. Impact of Preoperative Erythropoietin on Allogeneic Blood Transfusions in Surgical Patients: Results From a Systematic Review and Meta-analysis. Anesth Analg. 2019 May;128(5):981-992. doi: 10.1213/ANE.0000000000004005. PMID 30649068
- [Background] Kei T, Mistry N, Curley G, Pavenski K, Shehata N, Tanzini RM, Gauthier MF, Thorpe K, Schweizer TA, Ward S, Mazer CD, Hare GMT. Efficacy and safety of erythropoietin and iron therapy to reduce red blood cell transfusion in surgical patients: a systematic review and meta-analysis. Can J Anaesth. 2019 Jun;66(6):716-731. doi: 10.1007/s12630-019-01351-6. Epub 2019 Mar 28. PMID 30924000
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Li MH, Bolshinsky V, Ismail H, Burbury K, Ho KM, Amin B, Heriot A, Riedel B. A cross-sectional survey of Australian anesthetists' and surgeons' perceptions of preoperative risk stratification and prehabilitation. Can J Anaesth. 2019 Apr;66(4):388-405. doi: 10.1007/s12630-019-01297-9. Epub 2019 Jan 28. PMID 30693438
- [Background] Marshall KM, Loeliger J, Nolte L, Kelaart A, Kiss NK. Prevalence of malnutrition and impact on clinical outcomes in cancer services: A comparison of two time points. Clin Nutr. 2019 Apr;38(2):644-651. doi: 10.1016/j.clnu.2018.04.007. Epub 2018 May 2. PMID 29789167
- [Background] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Background] Mazzola M, Bertoglio C, Boniardi M, Magistro C, De Martini P, Carnevali P, Morini L, Ferrari G. Frailty in major oncologic surgery of upper gastrointestinal tract: How to improve postoperative outcomes. Eur J Surg Oncol. 2017 Aug;43(8):1566-1571. doi: 10.1016/j.ejso.2017.06.006. Epub 2017 Jun 23. PMID 28669651
- [Background] McKenna NP, Bews KA, Al-Refaie WB, Colibaseanu DT, Pemberton JH, Cima RR, Habermann EB. Assessing Malnutrition Before Major Oncologic Surgery: One Size Does Not Fit All. J Am Coll Surg. 2020 Apr;230(4):451-460. doi: 10.1016/j.jamcollsurg.2019.12.034. Epub 2020 Feb 26. PMID 32113029
- [Background] Minnella EM, Awasthi R, Loiselle SE, Agnihotram RV, Ferri LE, Carli F. Effect of Exercise and Nutrition Prehabilitation on Functional Capacity in Esophagogastric Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2018 Dec 1;153(12):1081-1089. doi: 10.1001/jamasurg.2018.1645. PMID 30193337
- [Background] Minnella EM, Bousquet-Dion G, Awasthi R, Scheede-Bergdahl C, Carli F. Multimodal prehabilitation improves functional capacity before and after colorectal surgery for cancer: a five-year research experience. Acta Oncol. 2017 Feb;56(2):295-300. doi: 10.1080/0284186X.2016.1268268. Epub 2017 Jan 12. PMID 28079430
- [Background] Ohkura Y, Ichikura K, Shindoh J, Ueno M, Udagawa H, Matsushima E. Relationship between psychological distress and health-related quality of life at each point of the treatment of esophageal cancer. Esophagus. 2020 Jul;17(3):312-322. doi: 10.1007/s10388-019-00710-y. Epub 2020 Jan 2. PMID 31897762
- [Background] Onstad MA, Schmandt RE, Lu KH. Addressing the Role of Obesity in Endometrial Cancer Risk, Prevention, and Treatment. J Clin Oncol. 2016 Dec 10;34(35):4225-4230. doi: 10.1200/JCO.2016.69.4638. Epub 2016 Nov 7. PMID 27903150
- [Background] Pal N, Broaddus RR, Urbauer DL, Balakrishnan N, Milbourne A, Schmeler KM, Meyer LA, Soliman PT, Lu KH, Ramirez PT, Ramondetta L, Bodurka DC, Westin SN. Treatment of Low-Risk Endometrial Cancer and Complex Atypical Hyperplasia With the Levonorgestrel-Releasing Intrauterine Device. Obstet Gynecol. 2018 Jan;131(1):109-116. doi: 10.1097/AOG.0000000000002390. PMID 29215513
- [Background] Papadia A, Ragni N, Salom EM. The impact of obesity on surgery in gynecological oncology: a review. Int J Gynecol Cancer. 2006 Mar-Apr;16(2):944-52. doi: 10.1111/j.1525-1438.2006.00577.x. PMID 16681794
- [Background] Rabischong B, Larrain D, Canis M, Le Bouedec G, Pomel C, Jardon K, Kwiatkowski F, Bourdel N, Achard JL, Dauplat J, Mage G. Long-term follow-up after laparoscopic management of endometrial cancer in the obese: a fifteen-year cohort study. J Minim Invasive Gynecol. 2011 Sep-Oct;18(5):589-96. doi: 10.1016/j.jmig.2011.05.015. Epub 2011 Jun 29. PMID 21719359
- [Background] Ramirez PT, Frumovitz M, Bodurka DC, Sun CC, Levenback C. Hormonal therapy for the management of grade 1 endometrial adenocarcinoma: a literature review. Gynecol Oncol. 2004 Oct;95(1):133-8. doi: 10.1016/j.ygyno.2004.06.045. PMID 15385122
- [Background] Schier R, Levett D, Riedel B. Prehabilitation: The next challenge for anaesthesia teams. Eur J Anaesthesiol. 2020 Apr;37(4):259-262. doi: 10.1097/EJA.0000000000001167. No abstract available. PMID 32073409
- [Background] Silver JK. Cancer prehabilitation and its role in improving health outcomes and reducing health care costs. Semin Oncol Nurs. 2015 Feb;31(1):13-30. doi: 10.1016/j.soncn.2014.11.003. Epub 2014 Dec 3. PMID 25636392
- [Background] Wei J, Zhang W, Feng L, Gao W. Comparison of fertility-sparing treatments in patients with early endometrial cancer and atypical complex hyperplasia: A meta-analysis and systematic review. Medicine (Baltimore). 2017 Sep;96(37):e8034. doi: 10.1097/MD.0000000000008034. PMID 28906392
- [Background] West MA, Loughney L, Lythgoe D, Barben CP, Sripadam R, Kemp GJ, Grocott MP, Jack S. Effect of prehabilitation on objectively measured physical fitness after neoadjuvant treatment in preoperative rectal cancer patients: a blinded interventional pilot study. Br J Anaesth. 2015 Feb;114(2):244-51. doi: 10.1093/bja/aeu318. Epub 2014 Oct 1. PMID 25274049